CLINICAL TRIAL: NCT07078253
Title: Improving Food Access in East Flatbush Through a Community Partner Coalition in New York City (NYC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-00432; UL1TR001445 (NIH)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Food Insecurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- East Flatbush community (Experimental): Produce grown by Brooklyn Grange and tailored to the East Flatbush community will be provided weekly for 20 week to enrolled study participants .
  Interventions: Other: Produce box program

INTERVENTIONS:
Other: Produce box program — Each week during the 20-week study period, participants will pick up a box of fresh vegetables. All produce will be provided to the participants at no cost as part of the client choice pantry program. Participants will take home approximately 6 different types of vegetables each week. Participants will choose which vegetables they want from a variety of options.

SUMMARY:
The objective of this research study is to implement and evaluate a food pantry pilot program to improve access to food and overall diet quality in East Flatbush. This will be achieved through the implementation of a tailored, client-choice food pantry pilot program. The pilot program will specifically offer locally grown produce.

DETAILED DESCRIPTION:
The objective of this study is to implement and evaluate a pilot intervention to improve access to food and overall diet quality in East Flatbush in Brooklyn, NY. This will be achieved through implementation of a tailored, client-choice pantry model pilot intervention among up to 100 individuals in which local, fresh produce is provided to participants on a weekly basis for 20 weeks. This project is a partnership between NYU and five community-based organizations (CBOs) and is the result of multi-year formative research with the partners and community. The pantry program will be evaluated using surveys and an objective measure of fruit and vegetable intake (i.e., skin carotenoid assessment via the Veggie Meter) at the start and end of the 20-week program. Through this pre-post evaluation, the investigators will assess the impact of the program on food security (primary outcome) as well as on fruit and vegetable intake and social connection (secondary outcomes). The findings will inform future implementations of client-choice pantry models by community-based organizations across New York City.

ELIGIBILITY:
Inclusion Criteria:

1. Adult at least 18 years old
2. Able to complete the surveys in English or Haitian Creole
3. Able to travel to Brooklyn Center for Quality Life in East Flatbush weekly to pick up the no-cost fresh vegetables
4. Willing and able to provide informed consent to participate in the study

Exclusion Criteria:

1) Those not meeting the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in the percent of individuals who report that they are low or very low food security households | Baseline, Week 20
  Outcome measure is assessed through a self-administered survey.

SECONDARY OUTCOMES:
Change in carotenoid levels | Baseline, Week 20
  The Veggie Meter is a portable electronic device that uses a light scan of the participant's finger to measure carotenoid levels, a validated marker of fruit and vegetable intake across diverse populations.
Change in social cohesion | Baseline, Week 20
  Social cohesion will be self-reported using questions about the neighborhood and related social interactions

CONTACTS AND LOCATIONS:
Overall Officials: Madison N LeCroy, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD data will not be made available due to the following key reasons. First, the possibility of re-identification of participants if IPD were shared is more than minimal given the small sample size and community-based recruitment. Participants have expressed heightened concerns about data security, and thus the study team will take efforts to protect participants by restricting access to their IPD. Secondly, data-sharing de-identified IPD is not included in the study's consent form, and re-consenting enrolled participants with this added stipulation would not be feasible.